CLINICAL TRIAL: NCT00760331
Title: A Long Term Follow up of a Cohort of Children With TCF2 Mutation:Evolution of Endocrine and Renal Function
Brief Title: Long Term Follow up of a Cohort of Children With TCF2 Mutation:Evolution of Endocrine and Renal Function
Acronym: TCF2
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: I06026
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2015-02

CONDITIONS: Hepatocyte Nuclear Factor 1-beta
Keywords: HNF1B; TCF2; MODY-5; CAKUT; Anomaly of renal development
MeSH Terms: conditions — Prostate Cancer, Hereditary, 11; Cakut

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Anomalies of renal development are well know for patients treated for MODY-5 diabetes due to TCF2 mutation.A recent study confirms the existence of pediatric patients having TCF2 mutation but presenting renal anomalies alone.Endocrine and renal evolution of these patients is unknown.The aim of this study is to follow a cohort of patients with TCF2 mutation and initially presenting renal anomalies alone.

DETAILED DESCRIPTION:
Biologic analysis and renal ultrasonography once a year.

After puberty or before kidney transplantation

* Abdominal and pelvic MRI
* Intravenous Glucose Tolerance Test

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting an anomaly of renal development due to TCF2 mutation
* Age<18 years old

Exclusion Criteria:

* Anomaly of renal development without TCF2 mutation
* Age≥18 years old
* Parents or patients refusing to participate to the study

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: pediatric patients presenting an abnormality of kidney developmentdue to TCF2 mutation or deletion.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-06; Primary Completion 2033-07 (Estimated); Study Completion 2033-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent GUIGONIS, MD, Principal Investigator — University Hospital, Limoges
Locations (1):
- CHU de Limoges, Limoges, France